CLINICAL TRIAL: NCT06605742
Title: The Effectiveness of The Support and Counseling Program Based on the Roy Adaptation Model in Postmenopausal Women With Genitourinary Syndrome
Brief Title: The Effect of Counseling Based on the Roy Adaptation Model on Sexual Life and Quality of Life in Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Arzu AKDEMİR, Assistant Professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9199
Record Dates: First submitted 2023-05-22; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Genitourinary Syndrome of Menopause; Female; Postmenopause
Keywords: Genitourinary Syndrome in Menopause; Roy's Adaptation Model; Sexual Health; Quality of Life

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Experimental Design
Masking Description: In the single-blind method, subjects do not know which of the experimental or control groups they were selected and therefore which method was applied to them.The researcher knows the subjects selected for the experimental and control groups, and therefore which method was applied to which subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): A Support and Counseling Program Based on the Roy Adaptation Model and a training booklet were prepared for women diagnosed with MGS. During the study, 5 counseling sessions were held for 4 months (16 weeks).
  Interventions: Other: Consultancy
- Control Grup (Experimental): Women in the control group received routine care from the hospital. They filled out the scales at the first and last interviews. At the first interview, women in the control group were given an educational booklet.
  Interventions: Other: Consultancy

INTERVENTIONS:
Other: Consultancy — In the single-blind method, subjects do not know which of the experimental or control groups they were selected and therefore which method was applied to them.The researcher knows the subjects selected for the experimental and control groups, and therefore which method was applied to which subjects
  Other Names: Randomized Controlled Experimental Design

SUMMARY:
In this study, it was aimed to determine the effect of the support and counseling program based on the Roy Adaptation Model given to postmenopausal women with Genitourinary Syndrome on their sexual life and quality of life.

DETAILED DESCRIPTION:
Menopause, one of the important stages of a woman's life, is a gradual physiological change process that occurs simultaneously with age and developmental changes. According to the 2018 data of the Turkish Statistical Institute (TUIK), the average life expectancy for women is 80.7 years. With the prolongation of life expectancy, the number of women in the menopause period increases and women spend 1/3 of their lives in the menopause period. By 2030, the global population of menopausal women is expected to include 1.2 billion people. Menopause, which has an important place in a woman's life, has become one of the important women's health problems that should be considered in health service planning and delivery.

Menopause is defined as the permanent cessation of menstruation due to the absence of estrogen production from the ovaries. Estrogen deprivation that occurs during this period causes the emergence of various signs and symptoms that have a significant impact on quality of life, physical, mental and sexual health. As a result of hormonal deprivation and aging, the anatomy and function of the urogenital tissues are significantly affected and vulvovaginal atrophy may occur. The terms vulvovaginal atrophy and atrophic vaginitis were found to be insufficient to describe menopausal symptoms associated with changes in the vulva, vagina, and lower urinary tract due to estrogen deficiency, and the term "Genitourinary Syndrome in Menopause (MGS)" was developed for a more inclusive terminology.

MGS is defined as the sum of symptoms and signs associated with a decrease in estrogen and other sex steroids, including changes in the labia major/minor, clitoris, vestibule, vagina, urethra, and bladder. The prevalence of MGS is 70% and causes vaginal dryness, irritation/burning/itching in the vulva or vagina, decreased lubrication during sexual activity, dyspareunia, postcoidal bleeding, frequent urination, and urinary incontinence. Srisukho et al. (2019) conducted among Thai postmenopausal women, the most common symptoms were found to be nocturia (77.7%) and vaginal dryness (51.7%). Moral et al. (2018) found that postmenopausal women most commonly experience vaginal dryness (93.3%) and decreased lubrication in sexual activity (90.0%). Selvi et al. (2020) similarly found that postmenopausal women most commonly experienced vaginal dryness (66.2%), decreased lubrication (55.3%), urgency (54.8%) and urinary incontinence 39.2%. Although these complaints negatively affect the daily life activities, quality of life and sexual health of postmenopausal women, women do not share their complaints with health care providers and often believe that they are a natural part of aging. Only 6-7% of postmenopausal women are treated. MGS associated with menopause and aging is usually permanent, unlike menopausal symptoms that disappear from time to time, such as hot flashes, but most women have no knowledge of the causes and effects of this condition. In the Vaginal Health: Perceptions, Perceptions, and Attitudes (VIVA) survey, 55% of women with vaginal conditions reported experiencing symptoms for 3 years or more, and only a minority (4%) attributed their symptoms to MGS. Age, attitudes towards menopause, sexual activity, chronic diseases, biopsychosocial reasons affect the level of MGS-related problems and the rate of seeking treatment. Chua et al. (2017) in a study conducted in five European countries, the rate of referral to healthcare professionals with the complaint of MGS was found to be in Asia (25%), the United States (56%), and Europe (62%). MGS is an under-recognized medical problem by healthcare providers and under-reported by women. Therefore, recent research suggests that healthcare providers should be proactive in helping their patients explain symptoms related to MGS. Most women expect their healthcare providers to initiate conversations about MGS complaints. Several studies of women with self-reported, MGS symptoms have shown that poor MGS management may be the result of poor awareness, reluctance to seek timely medical advice, and lack of communication between healthcare professionals.

Early recognition of signs and symptoms of MGS, provision of communication tools to facilitate dialogue, development of patient-based education programs and individual counseling are the basic steps that will help women to protect their sexual health and quality of life.While preparing the consultancy program, its preparation in accordance with the conceptual and theoretical framework will facilitate the execution and monitoring of the service. In this respect, the Roy Adaptation Model (RAM) supports the adaptation process of women with MGS complaints. According to RAM, adaptation is a set of processes in which an individual responds to environmental changes or stimuli. RAM examines stimuli in three groups as both internal and external factors. focal stimuli; are the focal stimuli that directly cause the adaptive response to which the individual immediately responds. contextual stimuli; are all other stimuli that contribute to the effect of the focal stimulus. All stimuli that are not the direct cause of the behavior, but affect the behavior and can be measured. residual stimuli; They are stimuli that can affect the individual but cannot be measured objectively. The person may not be aware of this factor or the effect of the factor may not be observed. Stimuli from the internal and external environment, in turn, activate regulatory and cognition coping mechanisms that generate behavioral responses related to physiological, self-concept, role function, and interdependence. The response of the individual occurs as a result of the stimulus and the level of adaptation. As a result, the individual exhibits adaptive behavior that maintains its integrity or ineffective, negative behavior. If a person constantly adapts, the result is health, and if the coping mechanism is insufficient, the result is disease. The goal of nursing interventions in RAM is to increase adaptive responses in each of the four adaptive domains in health and disease states. According to Roy, the four adaptive domains are independent of each other; At the same time, they have an impressive and integrating feature. A change in any of these adaptive areas causes changes in other areas. Roy Adaptation Model considers healthy and sick individuals as a whole with their physiological, psychological and social aspects. The model's use of the method of recognizing the individual in all aspects facilitates nursing interventions.

RAM is widely used as a conceptual model to guide education, research, practice and knowledge development. Elmoneim et al. (2017) found that a training program based on the Roy Adaptation Model had a positive effect on sexual function and spousal support among women with total hysterectomy. In a study conducted with a group of women in the menopausal period, it was found that the Roy Adaptation Model guides the assessment of women's adaptation levels and facilitates the management of stimuli to promote their adaptation, providing a holistic approach to evaluate and analyze the menopausal transition. In this context, it can be said that providing consultancy in accordance with the RAM model will increase the effectiveness of the consultancy service.

There are a limited number of studies on the implementation of training and consultancy for MGS in our country. As a result, the need for education and counseling is inevitable when the prevalence of MGS and the negative effects of the complaints on women's quality of life and sexual life are considered. It is thought that the counseling program based on the Roy Adaptation Model to be given to women suffering from MGS will contribute to the quality of life and sexual life of women. The educational content to be created with this study will form a direction for future studies, and the materials (booklet, etc.) to be prepared will serve as a resource for health professionals. Visibility of the problem and awareness of MGS will be provided and it will guide future researches. This study will contribute to the literature by examining the effect of the Roy Adaptation Model-based counseling program given to women with MGS complaints on their sexual life and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 40-60
* Verbal communication established
* Having an active sex life
* No menstruation for at least 1 year
* It has been determined that she has entered menopause with the hormone value in the blood (FSH above 25).
* Women who agree to participate in the study will be included in the sample group.

Exclusion Criteria:

* Those with advanced prolapse
* Those with Urinary Incontinence
* Those with systemic HRT
* Those who have neurological or psychiatric disorders, use antidepressants and derivatives
* Women who do not agree to participate in the research will be excluded from the study.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postmenopausal women diagnosed with Genitourinary Syndrome in Menopause
Enrollment: 92 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Sexual functions | 5 months
  FSFI (Female Sexual Function Index) was used to evaluate sexual function. FSFI is a 19-item scale developed by Rosen et al. (2000) to evaluate female sexual function. Turkish validity and reliability study was conducted by Öksüz and Malhan in 2005. FSFI evaluates sexual function or problems involving the last four weeks. A minimum raw score of 4 and a maximum raw score of 95 can be obtained from the scale. After scoring by multiplying the effect coefficients determined for the sub-dimensions, the lowest score is 2 and the highest score is 36, and as the score increases, sexual functions are maintained more adequately.
The quality of life of postmenopausal women | 5 months
  The Menopause Specific Quality of Life Questionnaire- MENQOL was used to assess quality of life. MENQOL is a self-administered tool developed by Hilditch et al. (1996) to assess the quality of life of menopausal women. The Turkish validity and reliability study of the scale was conducted by Kharbouch and Şahin. In MENQOL, each question item is scored between 1-8 points. A score of 1 indicates that there is no problem related to that issue, a score of 2 indicates that the issue exists but is not disturbing at all, and scores between 3-8 indicate the severity of the existing problem. A low score indicates a high quality of life in women.
Vaginal symptoms | 5 months
  The International Consultation on Incontinence Questionnare-Vaginal Symptoms (ICIQVS) was used to evaluate vaginal symptoms. The ICIQ-VS scale was developed by Price et al. in 2006. Turkish validity and reliability study was conducted by Rüstemoğlu and Aslan (2021). The ICIQ-VS scale consists of 14 questions, 25 items with sub-questions, and 3 sub-dimensions (vaginal symptoms, sexual issues and quality of life).
Depression | 5 months
  Beck Depression Scale was used to evaluate depression. It was developed by Beck et al. The Turkish validity and reliability study was conducted by Hisli in 1989. The BDI consists of 21 items assessing the severity of depression. The total score for the whole scale ranges from 0 to 63 points. The degree of depression is indicated by the total score

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Msc Akdemir, Study Director — İstanbul University-Cerrrahpaşa
Locations (1):
- İstanbul University-Cerrrahpaşa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Aliei MM.,Ghelichkhani F., Pakghohar M., Abadi MMM.,2016, Effectiveness of a sex education program on sexual function in postmenopausal women with sexual dysfunction: A randomized tria,In: Payesh, Vol 15, Iss 2, Pp 181-192.
- [Background] Angelou K, Grigoriadis T, Diakosavvas M, Zacharakis D, Athanasiou S. The Genitourinary Syndrome of Menopause: An Overview of the Recent Data. Cureus. 2020 Apr 8;12(4):e7586. doi: 10.7759/cureus.7586. PMID 32399320
- [Background] ACOG Practice Bulletin No. 141: management of menopausal symptoms. Obstet Gynecol. 2014 Jan;123(1):202-216. doi: 10.1097/01.AOG.0000441353.20693.78. PMID 24463691